Assessment of Safety of Air Travel in Patients with Birt-Hogg-Dube Syndrome

NCT03040115

Statistical analysis plan

Document date: August 5, 2015

The rate of pneumothorax will be estimated as a percentage of the number of flights taken. Because retrospective distinction between persistent and recurrent pneumothorax can be problematic, all ipsilateral pneumothoraces reported within the same month will be considered as one episode. If a given pneumothorax was treated with more than one intervention (e.g., chest tube followed by chemical pleurodesis followed by surgical pleurodesis), the most aggressive intervention (e.g., in this case, surgical pleurodesis) will be listed as the treatment of record for that event. For the purpose of our study, a pneumothorax that happened either during an air flight or within 24 hours after a flight will be defined as flight-related pneumothorax. We will compare other disease and patient characteristics to try to determine factors associated with an increased risk of in-flight pneumothorax. Statistical significance will be set at P value of 0.05 and determined by the chi-square test and the z-statistic, as appropriate. All analyses will be done by using SAS for Windows, version 9.4, Cary, NC.